CLINICAL TRIAL: NCT01192503
Title: Safety and Efficacy of Rasagiline in Restless Legs Syndrome
Acronym: RAS-RLS
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: University of Virginia (Other)
Collaborators: Teva Neuroscience, Inc. (Industry)
Responsible Party: Principal Investigator, Colleen P Harman, Project Manager, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14630
Record Dates: First submitted 2010-08-23; First posted 2010-09-01 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-02

CONDITIONS: Restless Legs Syndrome
Keywords: Restless Legs Syndrome; rasagiline; futility
MeSH Terms: conditions — Restless Legs Syndrome | interventions — rasagiline; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- rasagiline (Active Comparator)
  Interventions: Drug: rasagiline
- placebo (sugar pill) (Placebo Comparator)
  Interventions: Drug: placebo (sugar pill)

INTERVENTIONS:
Drug: rasagiline — 1mg (2 tablets of 0.5mg) at bedtime taken by mouth for 12 weeks
  Other Names: Azilect
  Arms: rasagiline
Drug: placebo (sugar pill) — 1mg (2 tablets of 0.5mg) taken at bedtime by mouth for 12 weeks
  Arms: placebo (sugar pill)

SUMMARY:
The purpose of this study is to find out if rasagiline improves RLS symptoms. We also want to make sure rasagiline is safe to give people with RLS.

DETAILED DESCRIPTION:
The primary objective is to determine if rasagiline, at a dosage of 1mg/day, is non-futile for the treatment of RLS, as measured by the International RLS Study Group Rating Scale (IRLS). The primary outcome variable will be the change in IRLS from baseline to Week 12.

The secondary objectives are to determine if rasagiline, at a dosage of 1mg/day, is safe and well-tolerated in participants with RLS. Also, to determine if rasagiline improves measures of global clinical change, sleep quality, excessive sleepiness, quality of life, or depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Men and women at least 18 years of age, capable of providing informed consent
* Diagnosed with idiopathic RLS, defined as meeting the International RLS Study Group diagnostic criteria without evidence for secondary causes of RLS
* Moderate or severe symptoms, defined as a score of 15 or greater on the International RLS Study Group Rating Scale (IRLS)
* Not currently receiving treatment for RLS. A 30-day washout period will be required for participants on dopamine agonists or other therapies. Stable doses of iron supplementation will be allowed
* On a stable dose of the following antidepressants, for at least 30 days prior to baseline visit:

  * Amitriptyline, up to 50mg/day
  * Trazodone, up to 100mg/day
  * Citalopram, up to 20mg/day
  * Escitalopram, up to 10mg/day
  * Paroxetine, up to 30mg/day
  * Sertraline, up to 100mg/day
* Female subjects must not be of childbearing potential or must agree to use of contraception for duration of study

Exclusion Criteria:

* Signs consistent with a secondary cause of RLS:
* History of initial unresponsiveness to dopaminergic RLS treatment despite adequate dose of initial therapy
* Use of another MAO inhibitor within 30 days of baseline visit
* Allergy or adverse reaction to rasagiline
* Prior adverse reaction to tyramine-containing foods
* Use of meperidine or other opiates within 30 days of the baseline visit
* Use of benzodiazepines within 30 days of the baseline visit
* Use of antidepressants, including TCAs, SSRIs, and SNRIs, except for those permitted as listed above
* Use of other drugs or supplements contraindicated with rasagiline, including St. John's wort, mirtazapine, cyclobenzaprine, dextromethorphan, cold products that contain ephedrine, pseudoephedrine
* Scheduled to undergo elective surgery during the course of the study
* Active medical or psychiatric illness that requires changes to treatment during the course of the study or jeopardize the subject's ability to remain in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2010-09; Primary Completion 2012-06 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Change in International Restless Legs Syndrome Study Group Rating Scale (IRLS) score from Baseline to Week 12 | Screening, Baseline, Week 6, Week 12
  The IRLS is a 10-question scale that contains questions about both the frequency and severity of RLS symptoms, as well as secondary aspects such as sleep quality and daytime tiredness.

SECONDARY OUTCOMES:
Tolerability (ability to complete study on assigned dosage) | 12 weeks
Adverse events | 12 weeks
Change in Beck Depression Inventory from Baseline to Week 12 | Baseline, Week 6, Week 12
Change in Clinical Global Impression - Change from Baseline to Weeks 12 | Baseline, Week 6, Week 12
Change in Medical Outcome Study Sleep Scale from Baseline to Week 12 | Baseline, Week 6, Week 12
Change in Johns Hopkins Restless Legs Syndrome Quality of Life Questionnaire from Baseline to Week 12 | Baseline, week 6, Week 12
Change in Epworth Sleepiness Scale from Baseline to Week 12 | Baseline, Week 6, Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Tiffini S Voss, MD, Principal Investigator — University of Virginia, Department of Neurology; Bernad Ravina, MD. MSCE, Principal Investigator — University of Rochester, Movement and Inherited Neurological Disorders Unit
Locations (8):
- United States (8):
  - Advent Research, Pinellas Park, Florida
  - Medical College of Georgia Movements Disorders Program, Augusta, Georgia
  - Northwestern University PD and Movement Disorders Center, Chicago, Illinois
  - Atlantic Neuroscience Institute Overlook Hospital, Summit, New Jersey
  - SUNY- Buffalo Jacobs Neurological Institute, Buffalo, New York
  - Cleveland Clinic Sleep Disorders Center, Cleveland, Ohio
  - University of Pennsylvania Sleep Center, Philadelphia, Pennsylvania
  - Charlottesville Medical Research, Charlottesville, Virginia